CLINICAL TRIAL: NCT00861068
Title: A Multi-Centre, Randomized, Double-Blind, Placebo Controlled Pilot Trial to Assess the Efficacy, Safety, and Tolerability of SPM 927 in Subjects With Postherpetic Neuralgia (PHN).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Study Director, UCB
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP0655
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Postherpetic Neuralgia
Keywords: Lacosamide, Vimpat®
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — 2-(acetylamino)-3-methoxy-N-(phenylmethyl)-, (2R)-; Lacosamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: SPM927/Lacosamide
- 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SPM927/Lacosamide — SPM927 (film-coated tablets, 25/50/100mg per tablet), dosage up to 600mg/day, intake in the morning and in the evening, intake for 11 weeks
  Arms: 1
Other: Placebo — Placebo tablets two times a day for 10 weeks
  Other Names: SPM927; Lacosamide; Vimpat®
  Arms: 2

SUMMARY:
The objective of the trial is to investigate the analgesic efficacy of SPM 927 in subjects with moderate to severe neuropathic pain due to Postherpetic Neuralgia (PHN)

ELIGIBILITY:
Inclusion Criteria:

* Subject has clinically diagnosed painful postherpetic neuralgia present at least six months after healing of a herpes zoster skin rash and has at least one form of allodynia
* Subject must have at least moderate pain (mean pain intensity ≥ 4 out of 10 during the baseline week on Likert scale).

Exclusion Criteria:

* Subject has other conditions that cause pain at least as severe as the postherpetic neuralgia.
* Subject has had any surgical treatment or any neurolytic injections for PHN
* Subject has clinically significant ECG and laboratory abnormalities.
* Subject is receiving treatment with anti-epileptic drugs (AEDs), muscle relaxants, mexiletine, topical analgesics, antidepressants, opioids, non-steroidal anti-inflammatory drugs (NSAIDs), paracetamol, benzodiazepines, and antiviral agents.
* Subject has liver function tests (AST, ALT, alkaline phosphatase, total bilirubin and GGT out of the reference range) > 1,5 x ULN (upper limit of normal) at visit 1
* Subject has serum creatinine ≥ 2 times the upper limit of reference range at Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2002-02; Primary Completion 2002-12 (Actual); Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Within-subject change in average daily pain score (Likert categorical scale) from the baseline week to the maintenance phase | Daily Assessments via patient diary and during patient's visit at the site

SECONDARY OUTCOMES:
Different qualities of pain due to PHN, sleep and activity (daily assessment during entire trial participation) | Daily assessment during entire trial participation including visits at the site
Investigate the tolerability and safety of SPM927 (assessments and reporting during entire trial participation). | Daily assessment during entire trial participation including visits at the site
To examine the pharmacokinetics of SPM927 (assessment at all site visits during entire trial participation) | Daily assessment during entire trial participation including visits at the site

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)